CLINICAL TRIAL: NCT00299052
Title: The Efficacy of Demineralized Bone Matrix and Autogenous Bone Graft in Accelerated Fracture Healing in Closed Tibia Fracture
Brief Title: Efficacy of DBM on Fractures of the Shinbone (Tibia)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Thomas Moore, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1272-2005; 3006
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Closed Fracture; Open Fracture
Keywords: Tibia; Fracture; DBM
MeSH Terms: conditions — Fractures, Closed; Fractures, Open; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Bone reamings with 5cc of DMB putty
  Interventions: Device: Grafton DBM
- B (Active Comparator): Bone reamings
  Interventions: Biological: Reamings

INTERVENTIONS:
Device: Grafton DBM — Grafton DBM will be mixed with bone reamings obtained during tibia IMN and place at the fracture site
  Arms: A
Biological: Reamings — Bone reamings obtained during tibia IMN will be placed at the fracture site
  Arms: B

SUMMARY:
The Tibia bone (shinbone) is located in the leg, itis the most frequently fractured bone in the body and has very poor blood supply because it is surrounded by skin and fat instead of muscle like the thighbone causing healing problems. Problems frequently found during the healing process are malunion (bone heals in the wrong place), nonunion (the bone never heals), and compartment syndrome (a big inflammation of muscle that causes compression of nerves and blood vessels) with necrosis (death) of tissue. Surgeons have tried to decrease these problems by using different surgical techniques and substances to accelerate healing. Substances frequently used in fractures are bone grafts. Bone grafts are normally obtained from the wrist or the hip bone, and sometimes can cause other complications varying from pain to infection. To avoid complications, investigators have used alternatives such as obtaining bone from donors. The donor bone grafts are carefully analyzed and cleaned to ensure they will not cause problems for the receiver. Bone obtained from donors is called Demineralized Bone Matrix (DBM). DBM has proved to be very effective in helping fractures to heal faster and we want to use it in patients with tibia fractures.

This study is important because DBM can improve the way tibia fractures are treated and could have the potential to decrease the time patients must stay in the hospital. DBM could improve healing time and diminish overall costs. Also, with the use of DBM plus reamings, patients will have fewer complications like pain and infection.

DETAILED DESCRIPTION:
Duration This study will last for 24 months.

Subject Recruitment

Inclusion criteria:

* Patients presenting diaphyseal tibia fractures.
* Patients older than 18 years old
* Patients that will undergo IM nailing as definitive treatment.

Exclusion criteria:

* Patients with systemic or bone infection.
* Patients with renal disease of any kind.

Location Emory Orthopedic Service at Grady Hospital

Background The tibia is the most common fractured bone. 14 It is also the bone with the higher incidence of open wounds because of the tibia proximity with the skin. 14 This bone is often in high risk of malunion, nonunion, infection, and other complications because of the tibia's precarious blood supply, and it is also associated with compartment syndrome in 1 to 9 % of cases. 10,14 Even though relatively new surgical procedures such as intramedullary nailing have increase the function recovery of this patients, still much is to be done to assure the proper evolution of the patients with tibia fractures. 10 It is important to find an adjuvant that will help with this recovery. It has been postulated that the use of bone graft could help in this process but there is more to be analyzed to drawn any definitively conclusion.

Tibia fractures are often part of the injuries in the polytrauma patient. Complicated fractures produced by trauma are often in the need for bone graft. Bone graft is usually obtained from the hip or the distal radius and the procedure is not exempt of complications such as pain, infection and increased hospitalization stay. In order to avoid these events, bone graft substitutes have been developed but most of them are expensive. 11 An example of this is bone morphogenic proteins (BMPs). BMPs have shown a high efficacy rate but cost wise, they could be prohibitive. 11 DBM could be a reasonable alternative and tentatively could have the same efficacy and less antigenic risks 5,9,11. Previous well designed studies have demonstrated the efficacy of demineralized bone matrix in fracture healing of non-unions, total joint osteolytic lesions, benign bone cysts and spine fusions.3-9,11-13 It has even proved it potential efficacy in restoring cartilage surface 7. The importance of this findings support the idea of using DBMs in other applications that could beneficiate the trauma patient.

DBMs are manufactured by different companies and they are available in different presentations. Most important, they vary also in their efficacy. The efficacy of a DBM depends mainly on it osteoconductivity and osteoinductivity 1,5. The differences in osteoconductivity and osteoinductivity between the available DBMs could represent a factor that limits the host's response to the graft 12. According to Louis-Ugbo et al, even the different presentations of DBM's could cause different host responses. 11 This is why it is very important to find a DBM that not only is highly effective, but also has the adequate presentation to be use in trauma fracture patients that require an acute treatment. In a study done by Cammisa et al they asseverate that the value of Grafton® is based upon not only the high osteoconductivity and osteoinductivity that the product presents, but also the fact that the gel formulation allows a mixture with allograft that helps to reach difficult graft sites 3. Other studies have shown that the putty presentation of Grafton® could be even higher in inductive properties 3. A previously done study at Grady Hospital conducted by our service reported an enhanced fracture healing in high energy tibial fractures treated with percutaneous injection of bone marrow with Grafton® acutely (reference to be inserted). Our experience support the hypothesis that Grafton® could be also valuable in the treatment of closed tibia diaphyseal fractures, with a smaller healing frame, decreased hospitalization time and early return to work.

Research Design

This study would randomize consecutive patients presenting closed tibia fractures into two groups:

* Group 1: Intramedullary (IM) rodding in standard fashion with the reamings.
* Group 2: IM rodding with intramedullary grafting with the reaming mixed with Grafton®.

We will randomize the patients using a list containing the patient research numbers and research groups. The research number will be assigned in order of presentation.

During the operative procedure, the patient will undergo the surgery as usual. In this particular surgery, the surgeon needs to follow the following steps:

1. An incision is made along the medial border of the patella tendon. This incision will be used to inset the nail into the intramedullary canal.10
2. The surgeon inserts an awl to through the bone metaphysis to access the medullary canal.10
3. A ball-tipped guide wire is now inserted into the tibial canal, passing across the fracture site.10
4. The canal is reamed in 0.5 mm increments. 10 The entry site is reamed until is wide enough to receive the nail.
5. After reaming, the ball-tipped guide is replaced by the permanent nail.
6. Proximal and distal screws are placed to avoid nail displacement
7. Incision wounds are closed and the patient is place in a splint.

The Grafton® mixture will be prepared by mixing the exceeding bone produced during reaming and the Putty Grafton® form. This preparation will be added during the surgery, before the permanent nail is situated. The mixture will be placed in the canal and positioned in the fracture site with the ball-tipped guide. Fluoroscopy images will be taken to assure the proper localization of the mixture. After this step, the permanent nail will be placed.

Both groups would undergo standard X-rays at appropriate times. Callus formation would be determined by standard radiographic (bridging callus measurement) and clinical evaluation (decreased pain at rest, with standing position and during ambulation)4. There will not be any alteration in length of stay or post-operative regimen. There will be scheduled post-op visits (one month, 6 weeks and 8 weeks) when X-rays of the tibia will be taken (AP, lateral and both oblique).

Visits

We will follow patients during their scheduled post-op visitis. They will be scheduled as follows:

Post op visit 1: 1 month after surgery Post op visit 2: 6 weeks after surgery Post op visit 3: 12 weeks after surgery Post op visit 4: 16 weeks after surgery Post op visit 5: 20 weeks after surgery. If necessary, we will include a visit 6 or 7 after 1 year or earlier according to the patient's needs.

Statistical Analysis Statistical analysis will be achieved by using Fisher's exact test 4. A P value <0.05 will be considered as statistically significant 4. For this pilot study we will enroll 30 patients, 15 per group, but we are planning to extend this number to 50 patients in a future, multicenter, randomized study. Using a two-sample t-test, the following analyses have been performed assuming a normal distribution of 2 samples with equal variances. If the mean time to fracture healing in group 1 is 42 days compared to 35 days for group 2, with a common standard deviation of 14 days for both groups, a sample size of 50 patients will be yield a significance level of .5 and power of .80.

Potential Risks Grafton® was associated with acute tubular necrosis in an animal study done with athymic rats 2,9. This study's authors suggested to restrain the use of DBM in children or patients with renal diseases 2,9. These findings have not been corroborated with any other study at the moment and there are some other points to be analyzed such as the associated materials used with Grafton®. In any case, we will not include patients with any type of renal disease or patients under the age of 18 years old in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting diaphyseal tibia fractures.

  * Patients older than 18 years old
  * Patients that will undergo IM nailing as definitive treatment.

Exclusion Criteria:

* Patients presenting diaphyseal tibia fractures.
* Patients older than 18 years old
* Patients that will undergo IM nailing as definitive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Fracture healing | Weeks 0-3, 4-6, 7-8, 12 and 16-24 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Moore, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States